CLINICAL TRIAL: NCT07148596
Title: Changes of Ciprofol Dosage and Bispectral Index Required for Loss of Consciousness in Patients of Different Ages: a Single-center, Prospective, Observational Study
Brief Title: Changes of Ciprofol Dosage and Bispectral Index Required for Loss of Consciousness in Patients of Different Ages
Status: Not yet recruiting | Type: Observational
Sponsor: General Hospital of Ningxia Medical University (Other)
Responsible Party: Sponsor
Other Study IDs: Yue Wen-2025-04
Record Dates: First submitted 2025-05-05; First posted 2025-08-29 (Actual); Last update posted 2025-08-29 (Actual); Status verified 2025-08

CONDITIONS: Ciprofol
Keywords: Bispectral index; Different ages; Loss of consciousness
MeSH Terms: conditions — Unconsciousness

STUDY DESIGN:
Observational Model: Other | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Other: It is an observational study without any intervention measures. — All patients will fast for 6 hours and will abstain from drinking for 2 hours preoperatively, with no premedication. Preoxygenation will be performed with an oxygen flow rate of 6 L/min. Ciprofol will be continuously infused via a micropump at a rate of 12 mg/kg/h. During preoxygenation with a facemask, if respiratory depression occurs during ciprofol infusion, assisted ventilation via facemask will be initiated. After LOC and completion of observation indices, the anesthesiologist may administer midazolam (1-3 mg), sufentanil (0.2-0.5 μg/kg), and rocuronium (0.3-0.6 mg/kg) sequentially based on the patient's age, physical condition, and BIS values to complete anesthesia induction. If hypotension (systolic blood pressure <90 mmHg or <80% of baseline) or bradycardia (heart rate <50 beats/min) occurs during induction, vasoactive agents such as ephedrine or atropine will be administered for management.

SUMMARY:
This study aims to explore dose requirements for loss of consciousness and bispectral index changes during general anesthesia induction with ciprofol in patients of different ages, providing a reference for its rational clinical application.

DETAILED DESCRIPTION:
Ciprofol, a novel gamma-aminobutyric acid (GABA) receptor agonist, is structurally modified from propofol by adding a cyclopropyl group to its side chain, forming an R-type chiral structure. This modification enhances its affinity for GABA receptors, resulting in faster onset, rapid metabolism, higher potency, reduced injection pain, and milder respiratory/circulatory suppression. Ciprofol exhibits good safety and tolerability, smooth and rapid induction, complete recovery, and low incidence of injection pain, making it a promising alternative to propofol. Age is a critical factor influencing general anesthesia and anesthetic drug responses. Age-related changes in organ function affect pharmacokinetics and pharmacodynamics, leading to variations in required drug doses and characteristic electroencephalogram changes. Therefore, this study aims to compare ciprofol doses and BIS changes during general anesthesia induction across age groups, offering reference and guidance for clinical medication.

ELIGIBILITY:
Inclusion Criteria:

* 1) The ASA classification I-II 2) BMI range: 18.5 < BMI ≤ 24.9 kg/m² 3) Scheduled for elective general anesthesia surgery 4) Signed informed consent by the patient or legal guardian

Exclusion Criteria:

* 1) Patients with central nervous system disorders or using medications affecting the central nervous system 2) Patients with cardiac, hepatic, pulmonary, or renal dysfunction 3) History of alcohol or drug abuse 4) Allergy to the study drug 5) Patients with hematologic or metabolic diseases 6) Participation in other drug clinical trials within the past 4 weeks 7) Refusal to participate in the study

Min Age: 3 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: A total of 120 patients scheduled for general anesthesia were selected according to inclusion/exclusion criteria, with balanced age distribution and equal gender allocation (60 males and 60 females).
Sampling Method: Probability Sample
Enrollment: 120 (Estimated)
Dates: Start 2025-09-01 (Estimated); Primary Completion 2025-12-01 (Estimated); Study Completion 2025-12-20 (Estimated)

PRIMARY OUTCOMES:
Ciprofol dosage | During anesthetic Induction
  Ciprofol dose required to achieve loss of consciousness. Ciprofol was continuously infused via a micropump at a rate of 12 mg/kg/h. The Modified Observer's Assessment of Alertness/Sedation (MOAA/S) scale and loss of eyelash reflex were used to assess sedation depth, with evaluations performed every 5 seconds. A MOAA/S score ≤1 and loss of eyelash reflex were defined as loss of consciousness (LOC).
Bispectral index | Baseline (Before surgery)
  Bispectral index before infusion, at loss of consciousness, and at 1 and 3 minutes post-loss.

SECONDARY OUTCOMES:
Mean arterial pressure (MAP) | up to 3 minutes
  MAP before infusion, at loss of consciousness, and at 1 and 3 minutes post-loss.
heart rate (HR) | up to 3 minutes
  HR before infusion, at loss of consciousness, and at 1 and 3 minutes post-loss.
SpO₂ | up to 3 minutes
  SpO₂ before infusion, at loss of consciousness, and at 1 and 3 minutes post-loss.
Incidence of adverse reactions including respiratory depression and injection pain | Baseline (Before surgery)
  Respiratory depression was defined as meeting any of the following criteria: respiratory rate <10 breaths/min, arterial oxygen saturation <90%, arterial partial pressure of carbon dioxide (PaCO₂) ≥50 mmHg, or apnea lasting ≥15 seconds. Injection pain is a subjective discomfort experienced by conscious patients during ciprofol infusion, diagnosed based on clinical manifestations and patient-reported complaints.

CONTACTS AND LOCATIONS:
Locations (1):
- General Hospital of Ningxia Medical University, Yinchuan, Ningxia, China

IPD SHARING:
Plan to Share IPD: No